CLINICAL TRIAL: NCT06196073
Title: The Effectiveness of Visceral Osteopathy in Functional Constipation: A Randomized Controlled Trial
Brief Title: Visceral Osteopathy in Functional Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Erhan KIZMAZ, Research assistant, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Constipation
Record Dates: First submitted 2023-12-23; First posted 2024-01-09 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Functional Constipation
Keywords: Functional constipatiton; Visceral; osteopathy
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Parallel two group which are equal
Who Masked: Outcomes Assessor
Masking Description: Sealed envelope method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visceral osteopathy and conservative treatment (Experimental): Osteoaptic manual treatment techniques
  Interventions: Other: Osteopathic manual therapy; Dietary Supplement: conservative treatment
- conservative treatment (Experimental): Nutritional supplements
  Interventions: Dietary Supplement: conservative treatment

INTERVENTIONS:
Other: Osteopathic manual therapy — Bilateral oscillation therapy to the T10-L2 region for the regulation of sympathetic tone, suboccipital release technique for the regulation of parasympathetic tone, sacrum mobilization, celiac, mesenteric superior and inferior ganglion mobilizations, colon peristalsis and ileocecal valve mobilization for the treatment of functional dysfunctions, ascending colon mobilization, transverse colon. mobilization, descending colon fascia mobilization and sigmoid colon mobilization, peritoneal mobilization
  Arms: Visceral osteopathy and conservative treatment
Dietary Supplement: conservative treatment — Nutritional recommendations and necessary nutritional supplements to facilitate digestion and defecation

SUMMARY:
It is a functional bowel disease characterized by excessive straining during defecation, infrequent defecation, and the feeling of incomplete evacuation. There are very few studies investigating the incidence and prevalence of functional constipation.Non-pharmacological treatment methods, including lifestyle changes, are primarily recommended for the treatment of constipation. The aim of the study is to examine the effects of visceral osteopathic approaches on individuals diagnosed with functional constipation and compare them with conventional methods.

DETAILED DESCRIPTION:
Non-pharmacological treatment methods, including lifestyle changes, are primarily recommended for the treatment of constipation. In cases where success is not achieved with this method, pharmacological agents, biofeedback and surgical treatment methods can be applied depending on the severity of constipation. Lifestyle changes include increasing fiber and fluid intake and regular physical activity Osteopathic manual therapy (OMT) is the examination and treatment of the function of the neuromusculoskeletal system anatomy using non-invasive, generally safe manual techniques to improve functional body mechanics such as joint range of motion, muscle tone, circulation, body fluid pressures and exchanges, and nerve impulses. OMT is used for autonomic system regulation, balancing pelvic muscle tone, increasing gastrointestinal motility, preventing myofascial limitations and increasing the pump effect of the diaphragm (5,6). The positive effects of OMT on the microbiome are available in the literature.

Alternative treatments are needed because the costs of combating constipation are high. Non-invasive interventions are especially gaining importance.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer individuals aged 18 and over
* Clinical diagnosis with functional constipation based on ROMA IV criteria

Exclusion Criteria:

* Clinical diagnosis of a gastrointestinal disease other than constipation,
* Undergone abdominal surgery in the last 6 months,
* Having abdominal aortic aneurysm, acute rectal bleeding, malignant mass in the GIS,
* Pregnancy or suspected of pregnancy,
* Cliniclal diagnosis of neurological disease that may cause constipation,
* Expreinced unexplained fever, Individuals with night sweats and weight loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-23 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Constipation severity scale | 5 minutes
  It is a scale that evaluates individuals' defecation frequency, intensity and difficulty during defecation. The scale includes 16 questions. It has 3 sub-dimensions: fecal obstruction, colon laziness and pain. The score range that can be obtained from the scale is 0-73. high scores indicate symptoms are severe.
Constipation Quality of Life Scale | 5 minutes
  This scale is a self-rating scale consisting of 28 items and subscales of "anxiety/anxiety" (11 items), "physical discomfort" (4 items), "psychosocial discomfort" (8 items), and "satisfaction" (5 items). Item scores of the five-point Likert-type scale vary between 1 and 5. While patients answered the first and fifth parts of the scale as "Not at all (1)", "Quite a bit (2)", "Somewhat (3)", "Quite a lot (4)" and "A lot (5)", the second, third, In the fourth and sixth sections, he was asked to choose the most suitable one among the options "Never (1)", "Rarely (2)", "Sometimes (3)", "Often (4)", "Always (5)". . The highest score that can be obtained from the scale is 140 and the lowest score is 28. It is thought that as the scores from the scale increase, the quality of life is negatively affected. There should be no unanswered questions for coding to be done.
Bristol Stool Scale | 5 minutes
  Bristol Stool Scale Bristol Stool Scale classifies human feces into 7 groups. The shape of the stool varies depending on the length of time it stays in the colon. Although not entirely scientific, this chart helps healthcare professionals better perceive stool patterns when making a diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Erhan Kızmaz, PhD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No